CLINICAL TRIAL: NCT02818647
Title: Comparison of Cold Dissection Technique and Needle Monopolar Electrocautery Tonsillectomy
Acronym: TONSIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Berke Ozucer, Otolaryngologist, Medical Doctor, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TONSIL
Record Dates: First submitted 2016-06-19; First posted 2016-06-30 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Tonsillitis; Tonsillectomy; Tonsillar Hypertrophy
Keywords: tonsillectomy; electrocautery; postoperative pain; visual analogue scale
MeSH Terms: conditions — Pain, Postoperative | interventions — Tonsillectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- COLD-DISSECTION (Active Comparator): Cold Dissection Technique
  Interventions: Procedure: Tonsillectomy
- HOT-DISSECTION (Active Comparator): Needle Electrocautery Dissection Technique
  Interventions: Procedure: Tonsillectomy

INTERVENTIONS:
Procedure: Tonsillectomy — Tonsillectomy is the name of the surgery where tonsils are removed via capsullary dissection. There are various techniques and its basically removing the tonsil from its tonsillary fossa and conducting hemostasis with various equipments.

SUMMARY:
Patients 13-years-or older who undergo tonsillectomy operation (without another additional surgery) will be enrolled in the study. Randomly, one side is going to be operated with conventional cold-knife technique and hemostasis will be maintained with bipolar diathermy (25-30w). Contralateral tonsil is going to be operated with needle-tip monopolar electrocautery (10-12w) at Blend 1 mode and hemostasis will also be maintained with needle-tip monopolar cautery. Postoperative tonsillar fossa healing and pain is going to be evaluated for both sides separately with Visual Analogue Scale. All operations are going to be performed by a single surgeon and all evaluations are going to be carried out by another surgeon in a totally blinded fashion to avoid possible bias.

DETAILED DESCRIPTION:
Comparison of cold and hot tonsillectomy carried out with needle-point tip monopolar electrocautery: a prospective, randomized, blinded, controlled (paired design) : A Randomized Clinical Trial

Tonsillectomy surgery techniques are basically divided into cold steel knife dissection and other (hot) techniques where surgeons use electrocautery and other contemporary technological devices. Pros / cons of hot and cold techniques have been long researched in the literature. Parameters are: cost, postoperative bleeding rate, postoperative pain. (Leinbach RF) Latest research proved that monopolar electrocautery (EC) is ideal when cost/postoperative bleeding rate ratio is concerned. (Cunningham LC) Although EC presents as a viable option, hot techniques - although providing good advantages - result with a more painful postoperative period. Trade-off with electrosurgery is the heat generated to cut/coagulate the tissue also causes a variable amount of tissue necrosis consequent to thermal injury. This pain is associated with the thermal injury and consequent tissue necrosis. (Hetzler D) Needle electrocautery tips are thinner compared to conventional bovie tip. Their surface area is smaller and according to the study carried out by Farnworth et al. (Farnworth TK) cause reduced thermal injury compared to conventional blade tip.

The investigators' aim in this study is to compare cold-knife dissection + bipolar diathermy tonsillectomy with needle tip EC monopolar cautery. Study design was prospective, randomised, single-blinded and controlled (paired). Either right tonsil was operated with standard-needle electrocautery, contralateral side was operated with cold-technique; or vice-versa. Which side received which treatment was randomly assigned (Aksoy F)

Surgical Technique

Both tonsils were injected with lidocaine and epinephrine infiltration to anterior tonsillar plica before the operation. All surgeries were performed by the primary investigator (BO) under x2.5 loupes. Force 2 Electrosurgical Generator (The Valley Lab, Boulder,CO) was used to power both the monopolar and bipolar electrocautery. Bipolar cautery was used (25-30 Watts) in accordance with the literature. Monopolar electrocautery settings were adjusted to 'Blend 1' which is a summation of the coagluation and cutting waveforms (75% cutting, 25% coagulation). Cut power was adjusted to 10W, whereas coagulation power was set to 12 Watts.

Results and Evaluations

Postoperative tonsillar fossa healing and pain is going to be evaluated for both sides separately with Visual Analogue Scale. All operations are going to be performed by a single investigator and all evaluations are going to be carried out by another investigator in a totally blinded fashion to avoid possible bias. These evaluations are going to be carried out for 10 postoperative days. Tonsillar fossa healing will be evaluated according to scale reported by Magdy EA et al. on first, fifth and tenth postoperative day (Magdy EA). Patients will evaluate their pain 10 (maximum) , 0 (none) based on a Visual Analogue Scale. Results will be calculated as (mean+-SD) and compared statistically for significance with SPSS.

Discussion

A finer tip can give greater precision in dissection and can also affect the dispersion characteristics of the energy used to perform the dissection. The implication of this for tonsillectomy is that greater precision in dissecting the tonsil from the underlying muscle can potentially lead to less post-operative discomfort.

For those surgeons who choose to use an electrocautery technique for tonsillectomy, the greater precision of the needle-tip EC may enhance the results.

ELIGIBILITY:
Inclusion Criteria:

* 13-years old and older
* Informed consent
* Isolated tonsillectomy (without adenoidectomy, OSAS surgery etc )
* Tonsillar hypertrophy

Exclusion Criteria:

* Malignancy suspicion
* Additional simultaneous surgeries (adenoidectomy, OSAS etc)

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change of postoperative Pain | Postoperative first 10 days
  Visual Analogue Scale will be used to evaluate the change in postoperative pain

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziosmanpasa Taksim Research and Education Hospital, Department of Otorhinolaryngology, Istanbul, Gaziosmanpasa
  - Gaziosmanpasa Taksim Research and Education Hospital,, Istanbul, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cunningham LC, Chio EG. Comparison of outcomes and cost in patients undergoing tonsillectomy with electrocautery and thermal welding. Am J Otolaryngol. 2015 Jan-Feb;36(1):20-3. doi: 10.1016/j.amjoto.2014.08.016. Epub 2014 Sep 2. PMID 25304999
- [Background] Aksoy F, Ozturan O, Veyseller B, Yildirim YS, Demirhan H. Comparison of radiofrequency and monopolar electrocautery tonsillectomy. J Laryngol Otol. 2010 Feb;124(2):180-4. doi: 10.1017/S0022215109991642. Epub 2009 Nov 30. PMID 19943988
- [Background] Farnworth TK, Beals SP, Manwaring KH, Trepeta RW. Comparison of skin necrosis in rats by using a new microneedle electrocautery, standard-size needle electrocautery, and the Shaw hemostatic scalpel. Ann Plast Surg. 1993 Aug;31(2):164-7. doi: 10.1097/00000637-199308000-00016. PMID 8215134
- [Background] Wexler DB. Recovery after tonsillectomy: electrodissection vs. sharp dissection techniques. Otolaryngol Head Neck Surg. 1996 Apr;114(4):576-81. doi: 10.1016/S0194-59989670249-8. PMID 8643267
- [Background] Leinbach RF, Markwell SJ, Colliver JA, Lin SY. Hot versus cold tonsillectomy: a systematic review of the literature. Otolaryngol Head Neck Surg. 2003 Oct;129(4):360-4. doi: 10.1016/S0194-59980300729-0. PMID 14574289
- [Background] Hetzler D. In reference to histologic assessment of thermal injury to tonsillectomy specimens: a comparison of electrocautery, coblation, harmonic scalpel, and tonsillotome. Laryngoscope. 2010 May;120(5):1077. doi: 10.1002/lary.20882. No abstract available. PMID 20422706
- [Background] Magdy EA, Elwany S, el-Daly AS, Abdel-Hadi M, Morshedy MA. Coblation tonsillectomy: a prospective, double-blind, randomised, clinical and histopathological comparison with dissection-ligation, monopolar electrocautery and laser tonsillectomies. J Laryngol Otol. 2008 Mar;122(3):282-90. doi: 10.1017/S002221510700093X. Epub 2007 Nov 26. PMID 18036277